CLINICAL TRIAL: NCT00728507
Title: A Phase II Randomized, Open-label Trial of a Rifapentine Plus Moxifloxacin-Based Regimen for Intensive Phase Treatment of Smear-Positive Pulmonary Tuberculosis
Brief Title: Rifapentine Plus Moxifloxacin for Treatment of Pulmonary Tuberculosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Johns Hopkins University (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0018
Record Dates: First submitted 2008-07-30; First posted 2008-08-05 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Moxifloxacin; Rifapentine
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Moxifloxacin; Pyrazinamide; Isoniazid; Rifampin; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Two months of isoniazid, rifapentine, pyrazinamide and moxifloxacin (HPZM) administered once daily. Pyridoxine (vitamin B6) will be given with each dose of isoniazid.
  Interventions: Drug: Rifapentine, Moxifloxacin, Pyrazinamide, Isoniazid
- 2 (Active Comparator): Two months of isoniazid, rifampin, pyrazinamide, and ethambutol (HRZE) administered once daily. Pyridoxine (vitamin B6) will be given with each dose of isoniazid.
  Interventions: Drug: Isoniazid, Rifampin, Pyrazinamide, Ethambutol

INTERVENTIONS:
Drug: Rifapentine, Moxifloxacin, Pyrazinamide, Isoniazid — Rifapentine:150mg tablets, dose = 300mg for subjects <= 45kg and 450mg for those >45kg by mouth once a day for 8 weeks; Moxifloxacin 400mg tablet by mouth once a day for 8 weeks, Isoniazid and Pyrazinamide per standard of care for TB treatment.
  Other Names: Priftin, Avelox
  Arms: 1
Drug: Isoniazid, Rifampin, Pyrazinamide, Ethambutol — Administered per standard of care for TB treatment
  Arms: 2

SUMMARY:
Although effective therapy for tuberculosis is available, TB continues to cause significant problems worldwide, and rates of multi-drug resistant (MDR) TB cases are on the rise. A major obstacle to the control of TB is poor adherence with lengthy (usually 6 months) and complicated treatment regimens. Incomplete TB treatment can lead to serious consequences such as increased severity of illness and death, prolonged infectiousness and transmission in the community, and the development of drug resistance. The development of new treatment strategies with more stronger drugs could lead to shorter and simpler regimens. A TB treatment regimen that allowed treatment duration to be meaningfully decreased would have important public health implications.

This trial will compare the effect and safety of a new oral regimen to that of the standard regimen for the first phase of treatment for pulmonary tuberculosis.

The experimental regimen will consist of the following:

* Two months of isoniazid, rifapentine, pyrazinamide and moxifloxacin (HPZM) administered once daily. Pyridoxine (vitamin B6) will be given with each dose of isoniazid.

The standard control intensive phase regimen will consist of the following:

* Two months of isoniazid, rifampin, pyrazinamide, and ethambutol (HRZE) administered once daily. Pyridoxine (vitamin B6) will be given with each dose of isoniazid.

Following intensive phase therapy (the study phase), all patients will be treated with a non-experimental continuation phase regimen.

In mice, the combination of Moxifloxacin and Rifapentine have cured the animals significantly faster than the standard regimen and this study will be the first step to see if the potential is also there in humans.

ELIGIBILITY:
Inclusion Criteria:

* Presumptive diagnosis of sputum smear-positive pulmonary TB.
* Age: ≥18 years
* Seven (7) or fewer days of multidrug therapy for TB disease in the preceding 6 months.
* Seven (7) or fewer days of fluoroquinolone therapy in the preceding 3 months.
* Documentation of HIV infection status.
* For HIV seropositive individuals, a CD4 T lymphocyte count of greater than or equal to 200 cells/mm3.
* Documentation of study baseline laboratory parameters done at, or ≤ 14 days prior to screening:

  * AST less than or equal to 2.5 times upper limit of normal.
  * Total bilirubin level less than 2.5 times upper limit of normal.
  * Creatinine level less than 2 times upper limit of normal.
  * Hemoglobin level of at least 8.0 g/dl.
  * Platelet count of at least 75,000 mm3.
  * Potassium level of at least 3.5.
  * Negative pregnancy test (women of childbearing potential).
* Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs).
* Male or nonpregnant, nonnursing female.
* Provision of informed consent.

Exclusion Criteria:

* CD4 count < 200 cells/cu mm.
* Presence of active AIDS-related opportunistic infection (other than TB) or active AIDS-related malignancy.
* Known intolerance to any of the study drugs.
* Concomitant disorders or conditions for which any of the study drugs is contraindicated. These include severe hepatic damage, acute liver disease of any cause, and acute uncontrolled gouty arthritis.
* Inability to take oral medication.
* Central nervous system TB.
* Pulmonary silicosis.
* Current or planned therapy, during study phase (intensive phase of TB treatment), with any one or more of the following drugs: quinidine, procainamide, amiodarone, sotalol, disopyramide, terfenadine, cisapride, erythromycin, clarithromycin, phenothiazines, haloperidol, olanzapine, ziprasidone, tricyclic antidepressants, chronic corticosteroids administered either orally or intravenously, chronic fluconazole,chronic itraconazole, chronic ketoconazole, oral or intravenous tacrolimus, oral or intravenous cyclosporine, HIV protease inhibitor, HIV non-nucleoside reverse transcriptase inhibitor.
* Concurrent severe and/or uncontrolled medical or psychiatric condition that, in the opinion of the investigator, could cause unacceptable safety risks or compromise compliance with the protocol.
* Unable or unwilling to receive directly observed therapy and/or adhere with follow-up (e.g. due to residence remote from the study site).
* Refusal of consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dorman, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- Brazil (3):
  - Centro de Referência Professor Hélio Fraga - ENSP - FIOCRUZ, Curicica, Rio de Janeiro
  - Posto de Saude Albert Sabin, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitario Clementio Fraga Filho, Rio de Janeiro

REFERENCES:
- [Background] Rosenthal IM, Williams K, Tyagi S, Peloquin CA, Vernon AA, Bishai WR, Grosset JH, Nuermberger EL. Potent twice-weekly rifapentine-containing regimens in murine tuberculosis. Am J Respir Crit Care Med. 2006 Jul 1;174(1):94-101. doi: 10.1164/rccm.200602-280OC. Epub 2006 Mar 30. PMID 16574936
- [Background] Nuermberger EL, Yoshimatsu T, Tyagi S, O'Brien RJ, Vernon AN, Chaisson RE, Bishai WR, Grosset JH. Moxifloxacin-containing regimen greatly reduces time to culture conversion in murine tuberculosis. Am J Respir Crit Care Med. 2004 Feb 1;169(3):421-6. doi: 10.1164/rccm.200310-1380OC. Epub 2003 Oct 24. PMID 14578218
- [Background] Nuermberger EL, Yoshimatsu T, Tyagi S, Williams K, Rosenthal I, O'Brien RJ, Vernon AA, Chaisson RE, Bishai WR, Grosset JH. Moxifloxacin-containing regimens of reduced duration produce a stable cure in murine tuberculosis. Am J Respir Crit Care Med. 2004 Nov 15;170(10):1131-4. doi: 10.1164/rccm.200407-885OC. Epub 2004 Aug 11. PMID 15306535
- [Derived] Conde MB, Mello FC, Duarte RS, Cavalcante SC, Rolla V, Dalcolmo M, Loredo C, Durovni B, Armstrong DT, Efron A, Barnes GL, Marzinke MA, Savic RM, Dooley KE, Cohn S, Moulton LH, Chaisson RE, Dorman SE. A Phase 2 Randomized Trial of a Rifapentine plus Moxifloxacin-Based Regimen for Treatment of Pulmonary Tuberculosis. PLoS One. 2016 May 9;11(5):e0154778. doi: 10.1371/journal.pone.0154778. eCollection 2016. PMID 27159505

RESULTS

PARTICIPANT FLOW:
Groups:
- HPZM: Two months of isoniazid, rifapentine, pyrazinamide and moxifloxacin (HPZM) administered once daily. Pyridoxine (vitamin B6) will be given with each dose of isoniazid.
  Rifapentine, Moxifloxacin, Pyrazinamide, Isoniazid: Rifapentine:150mg tablets, dose = 300mg for subjects <= 45kg and 450mg for those >45kg by mouth once a day for 8 weeks; Moxifloxacin 400mg tablet by mouth once a day for 8 weeks, Isoniazid and Pyrazinamide per standard of care for TB treatment.
- HRZE: Two months of isoniazid, rifampin, pyrazinamide, and ethambutol (HRZE) administered once daily. Pyridoxine (vitamin B6) will be given with each dose of isoniazid.
  Isoniazid, Rifampin, Pyrazinamide, Ethambutol: Administered per standard of care for TB treatment
Period: Overall Study
Arm/Group | HPZM | HRZE
Started | 62 | 59
Completed | 60 | 51
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPZM | HRZE | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [25 to 48] | 30 [24 to 45] | 32 [24 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 36 | 83
  Male | 15 | 23 | 38
Region of Enrollment [Number; unit: participants]
  Brazil | 62 | 59 | 121

OUTCOME MEASURES:

1. Primary Outcome: To Compare, by Treatment Group, the Percentage of Patients With a Negative Sputum Culture at the End of Intensive Phase Therapy.
Description: LJ culture conversion
Time Frame: Week 8
Population: modified intention to treat population
Measure: Number; unit: percentage of participants
Arm/Group | HPZM | HRZE
Number analyzed (Participants) | 60 | 51
percentage of participants | 78.3 | 84.3

2. Primary Outcome: To Compare the Safety and Tolerability of the 2 Intensive Phase Regimens.
Description: Study was prematurely terminated and data was not collected for this outcome measure.
Time Frame: Weekly or more frequent
Arm/Group | HPZM | HRZE
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | HPZM | HRZE
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 5/62 | 6/59
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HPZM (N=62) | HRZE (N=59)
flu-like syndrome (General disorders) | 2 | 0
change in visual refraction (Eye disorders) | 2 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 0
anemia (Blood and lymphatic system disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 0 | 1
hepatotoxicity (Hepatobiliary disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No